CLINICAL TRIAL: NCT05255406
Title: A Prospective, Single-arm, Phase 2 Clinical Trial of Furmonertinib as the First-line Treatment in EGFR-Mutant, PD-L1+ Patients With Locally Advanced or Metastatic NSCLC
Brief Title: Efficacy and Safety of Furmonertinib in EGFR-Mutant, PD-L1+ Patients With Locally Advanced or Metastatic NSCLC (FUTURE)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Huiyu, associate senior doctor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMTN-IIT-2021-001
Record Dates: First submitted 2022-02-16; First posted 2022-02-24 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aflutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Furmonertinib (Experimental): Furmonertinib (160mg)
  Interventions: Drug: Furmonertinib (160mg)

INTERVENTIONS:
Drug: Furmonertinib (160mg) — 160mg/day orally on a continuous dosing schedule. If subjects suffer from AEs, they can get declined dosage (80mg).
  Other Names: AST2818

SUMMARY:
The aim of this phase Ⅱ study is to evaluate the efficacy and safety of Furmonertinib in EGFR-Mutant, PD-L1+ Patients With Locally Advanced or Metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18 years old;
2. Locally advanced or metastatic non-squamous non-small cell lung cancer confirmed by histology or cytology (stage ⅢB-Ⅳ, according to the 8th Edition of the AJCC Staging system);
3. The tumour harbours one of the most common EGFR mutations (19del or L858R);
4. The programmed death-ligand 1 (PD-L1) tumoral expression is positive;
5. No previous systemic anti-tumor therapy for locally advanced or metastatic NSCLC;
6. According to RECIST 1.1, subjects have at least one measurable tumor lesion at baseline;
7. ECOG performance status score 0-2；
8. Subjects have voluntarily participated, signed and dated informed consent.

Exclusion Criteria:

1. Lung squamous carcinoma (including adenosquamous carcinoma and undifferentiated carcinoma) and small cell lung cancer;
2. Subjects have no measurable tumor lesion at baseline;
3. Subjects with spinal cord compression or symptomatic brain metastases;
4. Subjects are suitable for surgery;
5. Previous therapy with platinum-based chemotherapy, EGFR-TKIs, or anti-PD1/PD-L1 agents;
6. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT)>2.5 × ULN, or serum total bilirubin (TBIL)>1.5 × ULN, or Cr>1.0×ULN;
7. Absolute value of neutrophil (ANC)<1.5 × 109/L, or platelet (PLT) count<75 × 109/L, or hemoglobin (HGB)<90 g/L;
8. Any of the following disease within 12 months: myocardial infarction, severe/unstable stenocardia, coronary/peripheral artery bypass grafting, symptomatic congestive heart failure, or cerebrovascular accident;
9. Women who are pregnancy or lactation, or fertile but not using contraception;
10. Suffering from other serious acute or chronic physical or mental problems;
11. Subjects who are considered ineligible for the study for other reasons according to the investigator's assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
One-year Progression Free Survival Rate | One year after inclusion
  Percentage of subjects still alive and progression free one year after inclusion in the study.

SECONDARY OUTCOMES:
One-year Overall Survival Rate | one year after inclusion
  Percentage of subjects still alive one year after inclusion in the study.
Progression Free Survival | Approximately 2 years following the first dose of study drugs
  The time from the first does of the study drugs to the progression of the disease or death for any reason.
Objective Response Rate | Approximately 2 years following the first dose of study drugs
  Proportion of subjects whose tumors were assessed as complete response(CR) or partial response(PR) according to RECIST 1.1.
Adverse Events | Until 28 days from the last dose of study drugs or initiation of a new anticancer treatment
  Number of participants with adverse events as a measure of safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Yu, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No